CLINICAL TRIAL: NCT01225770
Title: Effects of Gargling With Green Tea on Preventing Influenza Infection Among High School Students: A Randomized Clinical Study
Brief Title: Gargling With Green Tea for Prophylaxis of Influenza Infection in Teenagers
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Shizuoka (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CT2010001
Record Dates: First submitted 2010-10-19; First posted 2010-10-21 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Influenza Infection
Keywords: green tea; gargling; prophylaxis; influenza; Respiratory Tract Infections; high school students
MeSH Terms: conditions — Influenza, Human; Respiratory Tract Infections | interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Green tea (Experimental): Gargling with green tea
  Interventions: Dietary Supplement: green tea
- water (Active Comparator): Gargling with water
  Interventions: Dietary Supplement: green tea

INTERVENTIONS:
Dietary Supplement: green tea — Gargling three times daily for 90 days

SUMMARY:
Experimental and clinical studies in adults have reported that green tea catechins prevent influenza infection. In this clinical randomized study, the investigators aimed to determine the effects of gargling with green tea on the prophylaxis of influenza infection among high school teenagers.

DETAILED DESCRIPTION:
Influenza infection is the principal cause of acute respiratory illnesses and occurs in epidemic or pandemic worldwide. It spreads easily among high school students and from them to the rest of the community; therefore the prevention of influenza is very important.

Experimental studies have revealed that some components of green tea can prevent influenza infection in vitro. In clinically, gargling with green tea catechins has been reported to have possibilities to preventing influenza infection in adults; however, little clinical evidence in teenagers has so far been existed. Based on this background, the investigators designed a randomized study to evaluate the clinical efficacy of gargling with green tea in preventing influenza infection among high school students.

ELIGIBILITY:
Inclusion Criteria:

* aged from 15 to 20 years
* obtained written informed consent from both the student and parent before participation
* possible to gargle during 90 days
* possible to fill in questionnaire

Exclusion Criteria:

* Possessing allergy to green tea
* Possessing history of influenza infection within 6 months before entering the study
* Possessing severe immune disease or whole body infection
* severe cardiac, respiratory, renal, or hepatic dysfunction
* diagnosed as inadequate to participate in the study by student doctor

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 640 (Estimated)
Dates: Start 2010-11; Primary Completion 2014-04 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
the incidence rates of influenza infection | Until 3 months gargling

SECONDARY OUTCOMES:
severity of influenza symptoms | until 3 months gargling
influenza-free time during the study period | until 3 months gargling
incidence of complications | until 3 months gargling
incidence rates of upper respiratory tract infections | until 3 months gargling
incidence of days of absence from school | until 3 months gargling
occurrence of the adverse events | until 3 months gargling

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Yamada, MD, PhD, Study Chair — University of Shizuoka
Locations (1):
- University of Shizuoka, Shizuoka, Shizuoka, Japan

REFERENCES:
- [Derived] Ide K, Yamada H, Matsushita K, Ito M, Nojiri K, Toyoizumi K, Matsumoto K, Sameshima Y. Effects of green tea gargling on the prevention of influenza infection in high school students: a randomized controlled study. PLoS One. 2014 May 16;9(5):e96373. doi: 10.1371/journal.pone.0096373. eCollection 2014. PMID 24836780